CLINICAL TRIAL: NCT01105052
Title: Cognitive Behavioral Therapy as Guided Self-help for Insomnia - a Randomized Controlled Trial
Brief Title: Self-help Cognitive Behavioral Therapy (CBT) for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stiftelsen Professor Bror Gadelius Minnesfond (Unknown)
Responsible Party: Mats Lekander, Karolinska Instutitet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008/23-31/4
Record Dates: First submitted 2010-04-12; First posted 2010-04-16 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Insomnia
Keywords: Insomnia; Co-morbid; CBT; Self-help; Bibliotherapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bibliotherapy (Active Comparator): A group receiving a self-help book to work on for six weeks with no therapist support.
  Interventions: Behavioral: Self-help CBT-I
- Bibliotherapy with support (Experimental): A group receiving a self-help book to work on for six weeks, together with brief weekly telephone calls (<15 minutes) from a therapist.
  Interventions: Behavioral: Self-help CBT-I
- Wait-list control group (No Intervention): This group receives no intervention until about five months after the two treatment groups, when participants in this group receive the self-help book without therapist support.

INTERVENTIONS:
Behavioral: Self-help CBT-I — Comparison between Bibliotherapy with and without support to a wait-list control group
  Arms: Bibliotherapy; Bibliotherapy with support

SUMMARY:
The purpose of this study is to investigate whether a self-help book for insomnia, with or without therapist support, can improve sleep and alleviate insomnia symptoms in individuals suffering from insomnia, also for persons presenting with different kinds of co-morbid problems.

DETAILED DESCRIPTION:
CBT has previously been identified as an effective treatment for insomnia. However, there is a lack of trained CBT-therapists, and self-help is beginning to prove useful for many areas of psychological distress. Earlier studies of different kinds of self-help (e.g. computer based and bibliotherapeutic) suggest that many patients do indeed benefit from self-help treatments for insomnia, but there is a need for independent replications. Also, most previous studies have had very strict inclusion criteria, such that for instance only individuals with primary insomnia and no co-morbid problems have been included. A general question in self-help is whether patients need therapist support to benefit from treatment, or if a book is enough to alleviate symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Diagnosis of Insomnia (Research Diagnostic Criteria)
* Access to computer
* Ability to read and write Swedish

Exclusion Criteria:

* Severe psychopathology (e.g. bipolar disorder, suicidality)
* Shift work

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Sleep diary | Six weeks after beginning of treatment
  Daily self-observation of sleeping behaviours used to calculate Total Sleep Time, Wake After Sleep Onset, Sleep Onset Latency, Sleep Efficiency, and gagues Sleep Quality, Daytime Ratings, Daytime Fatique and Bedtime Stress.
Sleep diary | 5 months after beginning of treatment (i.e. about three months after the end of treatment)
  Daily self-observation of sleeping behaviours used to calculate Total Sleep Time, Wake After Sleep Onset, Sleep Onset Latency, Sleep Efficiency, and gagues Sleep Quality, Daytime Ratings, Daytime Fatique and Bedtime Stress.
Sleep diary | 15 months after the end of treatment
  Daily self-observation of sleeping behaviours used to calculate Total Sleep Time, Wake After Sleep Onset, Sleep Onset Latency, Sleep Efficiency, and gagues Sleep Quality, Daytime Ratings, Daytime Fatique and Bedtime Stress.

SECONDARY OUTCOMES:
Insomnia Severity Index | Six weeks after beginning of treatment
  7-item patient-reported outcome assessing the severity of initial, middle and late insomnia; sleep satisfaction; interference of insomnia with daytime functioning; noticeability of sleep problems by others; and distress about sleep difficulties. A 5-point scale is used to rate each item, yielding a total score of 0 to 28. Higher score indicates more severe insomnia within 4 severity categories: absence of insomnia (score of 0-7); subthreshold insomnia (8-14); moderate insomnia (15-21) and severe insomnia (22-28).
Insomnia Severity Index | 5 months after beginning of treatment (i.e. about three months after the end of treatment)
  7-item patient-reported outcome assessing the severity of initial, middle and late insomnia; sleep satisfaction; interference of insomnia with daytime functioning; noticeability of sleep problems by others; and distress about sleep difficulties. A 5-point scale is used to rate each item, yielding a total score of 0 to 28. Higher score indicates more severe insomnia within 4 severity categories: absence of insomnia (score of 0-7); subthreshold insomnia (8-14); moderate insomnia (15-21) and severe insomnia (22-28).
Insomnia Severity Index | 15 months after the end of treatment
  7-item patient-reported outcome assessing the severity of initial, middle and late insomnia; sleep satisfaction; interference of insomnia with daytime functioning; noticeability of sleep problems by others; and distress about sleep difficulties. A 5-point scale is used to rate each item, yielding a total score of 0 to 28. Higher score indicates more severe insomnia within 4 severity categories: absence of insomnia (score of 0-7); subthreshold insomnia (8-14); moderate insomnia (15-21) and severe insomnia (22-28).

CONTACTS AND LOCATIONS:
Overall Officials: Mats Lekander, Ass prof, Study Chair — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Kraepelien M, Blom K, Forsell E, Hentati Isacsson N, Bjurner P, Morin CM, Jernelov S, Kaldo V. A very brief self-report scale for measuring insomnia severity using two items from the Insomnia Severity Index - development and validation in a clinical population. Sleep Med. 2021 May;81:365-374. doi: 10.1016/j.sleep.2021.03.003. Epub 2021 Mar 16. PMID 33813233
- [Derived] Jernelov S, Lekander M, Blom K, Rydh S, Ljotsson B, Axelsson J, Kaldo V. Efficacy of a behavioral self-help treatment with or without therapist guidance for co-morbid and primary insomnia--a randomized controlled trial. BMC Psychiatry. 2012 Jan 22;12:5. doi: 10.1186/1471-244X-12-5. PMID 22264332